CLINICAL TRIAL: NCT03070041
Title: Vauvamyönteisyysohjelman Vaikutus Imetykseen, Imetysohjaukseen ja Imetysasenteisiin / The Impact of Baby-friendly Hospital Initiative to Breastfeeding, Breastfeeding Counselling and Breastfeeding Attitudes
Brief Title: The Impact of Baby-friendly Hospital Initiative to Breastfeeding, Breastfeeding Counselling and Breastfeeding Attitudes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Hannakaisa Niela-Vilen, Post doc researcher, University of Turku
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Satavamy
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mothers and staff members (Experimental): The mothers who will give birth at the study hospital and all the staff members taking care about mothers and/or infants
  Interventions: Other: Baby-friendly Hospital Initiative

INTERVENTIONS:
Other: Baby-friendly Hospital Initiative — The intervention is Baby-friendly Hospital Initiative as described by WHO and UNICEF. The ten steps to successful breastfeeding will be implemented in the hospital.

SUMMARY:
The impact of Baby-friendly Hospital Initiative (BFHI) to breastfeeding, breastfeeding counselling and breastfeeding attitudes will be examined in Satakunta Central Hospital, Finland. The baseline measurement will be conducted before the implementation of BFHI in 2017 and second measurement will be conducted in 2019 after the certification process. Both staff members and breastfeeding mothers will be recruited in the study. The main outcomes are the duration of breastfeeding and breastfeeding attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Staff: All staff members taking care of mothers and/or infants in the hospital.
* Mothers: Mothers who have given birth in the study hospital during the data collection period.

Exclusion Criteria:

* Mothers:

  * who have given birth outside the hospital,
  * whose infant's condition is critical,
  * whose infants are transferred to another unit.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Duration of breastfeeding | Six months
  Duration of breastfeeding will be asked from the mother

SECONDARY OUTCOMES:
Breastfeeding attitude of the staff (questionnaire) | Two years
  Attitude will be measured with a structured questionnaire
Breastfeeding attitude of the mothers (questionnaire) | Four months
  Attitude will be measured with a structured and validated questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Satasairaala Central Hospital, Pori, Finland

IPD SHARING:
Plan to Share IPD: No